CLINICAL TRIAL: NCT06767475
Title: Effectiveness of Mindfulness-Based Intervention on Patient Reported Outcomes of Black Adult Cancer Survivors: A Community Faith-based Mindfulness Ministry (ComFaMM) Trial
Brief Title: Mindfulness-Based Stress Reduction to Improve Well-being in Black Adult Cancer Survivors, Community Faith-based Mindfulness Ministry
Acronym: ComFaMM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Floyd B. Willis, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MC240901; NCI-2024-10490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC240901 (Other: Mayo Clinic); 24-006322 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-01-02; First posted 2025-01-10 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Health Promotion; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I (MBSR) (Experimental): Patients participate in group discussions, exercises, and activities over no more than 8 hours for up to 3 sessions (up to 16 hours total).
  Interventions: Other: Health Promotion; Other: Questionnaire Administration
- Group II (control) (Active Comparator): Patients receive usual care on study.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Phase 0 (intervention development, pilot testing) (Experimental): INTERVENTION DEVELOPMENT: Participants may attend a focus group or a one-on-one interview over up to 60 minutes to gather insights of the cultural needs of Black adult cancer survivors.
  PILOT TESTING: Patients participate in a group discussion with exercises and activities on study.
  Interventions: Other: Discussion; Other: Health Promotion; Other: Interview; Other: Questionnaire Administration
- Phase 1 (MBSR) (Experimental): Patients participate in group discussions, exercises, and activities over no more than 8 hours for up to 3 sessions (up to 16 hours total) within 8 weeks.
  Interventions: Other: Health Promotion; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group II (control)
Other: Discussion — Attend a focus group
  Other Names: Discuss
  Arms: Phase 0 (intervention development, pilot testing)
Other: Health Promotion — Participate in group discussion with exercises and activities
  Other Names: Health Promotion (Salutogenesis); Health Promotion and Wellness; Mindfulness Health Promotion; Salutogenesis
  Arms: Group I (MBSR); Phase 0 (intervention development, pilot testing); Phase 1 (MBSR)
Other: Interview — Attend a one-on-one interview
  Arms: Phase 0 (intervention development, pilot testing)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the impact of a Mindfulness-Based Stress Reduction (MBSR) program adjusted to include Christian principles on well-being in Black adult cancer survivors. Cancer survivors face a unique set of challenges that includes not only physical but also mental and spiritual well-being. Concerns related to both diagnosis and treatment profoundly impact the quality of life of Black cancer survivors. Mindfulness-based interventions (MBIs) have been shown to be effective in improving psychological resilience, reducing anxiety, and enhancing the quality of life among cancer survivors. However, there is little research focusing on these interventions among Black adult cancer survivors. Research has shown that interventions that include cultural experiences, such as the role of religion, spirituality and faith, are more effective in maintaining psychological well-being in Black men. A MBSR program adjusted to include Christian principles may improve the well-being in Black adult cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop a culturally adapted Mindfulness-Based Stress Reduction (MBSR) intervention. (Phase 0) II. Pilot test the MBSR intervention to assess its feasibility, acceptability, and preliminary efficacy among a small group of participants. (Phase 0)

OUTLINE:

PHASE 0:

INTERVENTION DEVELOPMENT: Participants attend a focus group or a one-on-one interview over up to 60 minutes to gather insights of the cultural needs of Black adult cancer survivors.

PILOT TESTING: Patients participate in a group discussion with exercises and activities on study.

After completion of study intervention, patients are followed up at 3 months.

PHASE 1: Patients participate in group discussions, exercises, and activities over no more than 8 hours for up to 3 sessions (up to 16 hours total) within 8 weeks.

PHASE 2: Patients are randomized to 1 of 2 groups.

GROUP I (INTERVENTION): Patients participate in group discussions, exercises, and activities over no more than 8 hours for up to 3 sessions (up to 16 hours total).

GROUP II (CONTROL): Patients receive usual care on study.

After completion of study intervention, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PHASE 0 DEVELOPMENT: Adults aged 18 or older
* PHASE 0 DEVELOPMENT: Ability to speak, read and understand English
* PHASE 0 DEVELOPMENT: Individuals personally affected by cancer, either through their own diagnosis or that of a loved one
* PHASE 0 DEVELOPMENT: Self-identifies as Black or African American
* PHASE 0 DEVELOPMENT: Membership or affiliation with a faith-based organization
* PHASE 0 PILOT TESTING: Adults aged 18 or older
* PHASE 0 PILOT TESTING: History of a cancer diagnosis
* PHASE 0 PILOT TESTING: Meets National Cancer Institute (NCI) cancer survivor definition (a person is a survivor from the time of diagnosis until the end of life)
* PHASE 0 PILOT TESTING: Ability to physically attend live MBI and complete web-based surveys and assessments
* PHASE 0 PILOT TESTING: Ability to speak, read and understand English
* PHASE 1: Adults aged 18 or older
* PHASE 1: History of a cancer diagnosis
* PHASE 1: Meets NCI cancer survivor definition (a person is a survivor from the time of diagnosis until the end of life)
* PHASE 1: Ability to physically attend live MBI and complete web-based surveys and assessments
* PHASE 1: Ability to speak, read and understand English
* PHASE 2: Adults aged 18 or older
* PHASE 2: History of a cancer diagnosis
* PHASE 2: Meets NCI Cancer Survivor definition (a person is a survivor from the time of diagnosis until the end of life)
* PHASE 2: Ability to physically attend live MBI and complete web-based surveys and assessments
* PHASE 2: Ability to speak, read and understand English

Exclusion Criteria:

* PHASE 0 DEVELOPMENT: Does not meet the inclusion criteria
* PHASE 0 DEVELOPMENT: Unable or unwilling to participate in the recorded sessions
* PHASE 0 PILOT TESTING: Inability to attend and participate in MBI due to medical or psychological hardship
* PHASE 0 PILOT TESTING: Inability to speak, read and understand English
* PHASE 1: Inability to attend and participate in MBI due to medical or psychological hardship
* PHASE 1: Inability to speak, read and understand English
* PHASE 1: Participated in phase 0 of the study
* PHASE 2: Inability to attend and participate in MBI due to medical or psychological hardship
* PHASE 2: Inability to speak, read and understand English
* PHASE 2: Participated in phase 0 or phase 1 of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Spiritual well-being | Up to 3 months
  Will be measured by the change in scores on the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp-12). The FACIT-Sp-12a is a 12-item scale measuring spiritual well-being over the past 7 days. Responses are on a 5 point Likert-type scale (0=not at all; 1=a little bit, 2=somewhat; 3=quite a bit; 4=very much) with higher scores generally representing greater well-being

SECONDARY OUTCOMES:
Quality of life (QOL) | Up to 3 months
  Will be evaluated using changes in health related QOL patient reported outcomes responses. The World Health Organization Quality of Life Brief Version (WHOQOL-BREF) will be used to assess spiritual, religious or personal beliefs and how these beliefs have affected QOL including positive feelings, social support, self-esteem, pain, energy, work capacity, health and social care, and leisure activities. The WHOQOL-BREF is a 26-question instrument consisting of four domains. Each individual item of the WHOQOL-BREF is scored from 1-5 on a five-point ordinal scale.
Level of resilience - CD-RISC | Up to 3 months
  Will be measured by the Connor- Davidson Resilience Scale (CD-RISC). The CD-RISC is comprised of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience.
Level of resilience - RSA | Up to 3 months
  Will be measured by the Resilience Scale for Adults (RSA). The RSA examines intrapersonal and interpersonal protective factors presumed to facilitate adaptation to psychosocial adversities, as well as family and social protective factors of resilience. The RSA has 33 items; item-response ranges from one to seven; higher scores reflect higher levels of protective factors of resilience.
Personal spirituality and closeness with God | Up to 3 months
  Will be measured by change in spiritual variable adapted from Daily Spiritual Experience Scale (DSES) to assess perceived closeness to a higher power (God). The DSES is a 16-item self-report measure designed to assess ordinary experiences of connection with the transcendent in daily life. Responses are on a 6-point scale (many times a day; every day; most days; some days; once in a while; never) or 4-point scale (not at all; somewhat close; very close; as close as possible).
Overall assessment of the MBI and perception of MBI value | 3 months
  Will be assessed using the Was It Worth It (WIWI) questionnaire to determine changes in participants view on the worthiness of the intervention. Responses to the WIWI will capture participants' subjective evaluations of the intervention's impact. WIWI is a 3-item questionnaire with yes or no responses.

CONTACTS AND LOCATIONS:
Overall Officials: Floyd B. Willis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials